CLINICAL TRIAL: NCT02504775
Title: Single Blinded, Two-period, Two-treatment, Crossover, Randomized, Single Dose Bioequivalence Study of Two Oral Formulations With 500 mg of Paracetamol (Mejoral® 500 Tablets, Glaxosmithkline méxico s.a. De c.v. Vs. Tylenol® Caplets, Janssen Cilag de méxico, s. De r.l. De c.v.) in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study for Mejoral 500 Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 204779
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tylenol® Caplets, then Mejoral® 500 Tablets (Experimental): Participants will first receive one tablet [500 milligram (mg) of paracetamol] of Tylenol® Caplets, orally with 250 mL of water at room temperature, in a single dose, under minimum 10 h fasting. After a washout period of 72 h, they then will receive one tablet (500 mg of paracetamol) of Mejoral® 500 tablets, orally with 250 mL of water at room temperature, in a single dose, under minimum 10 h fasting.
  Interventions: Drug: Mejoral® 500 Tablets; Drug: Tylenol® Caplets
- Mejoral® 500 Tablets, then Tylenol® Caplets (Experimental): Participants will first receive one tablet (500 mg of paracetamol) of Mejoral® 500 tablets, orally with 250 mL of water at room temperature, in a single dose, under minimum 10 h fasting. After a washout period of 72 h, they then will receive one tablet (500 mg of paracetamol) of Tylenol® Caplets, orally with 250 mL of water at room temperature, in a single dose, under minimum 10 h fasting.
  Interventions: Drug: Mejoral® 500 Tablets; Drug: Tylenol® Caplets

INTERVENTIONS:
Drug: Mejoral® 500 Tablets — 500 mg tablet of paracetamol
Drug: Tylenol® Caplets — 500 mg tablet of paracetamol

SUMMARY:
This will be a monocentric, single blinded, randomized, single-dose, two-periods, two-sequence, crossover bioequivalence study of two oral formulations in healthy participants under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent
* Men and women between 18 to 55 years of age, with good state of health
* Participants' body mass index must be between 18.0 and 27.0
* Blood pressure (seated) up to 139 milliliters of mercury (mm/Hg) systolic and up to 89 mm/Hg diastolic, heart rate between 60 and 100 beats per minute and respiratory frequency between 14 and 20 breaths per minute
* The laboratory tests: Complete blood count with differential count, Chemical blood of 27 elements, Urinalysis, Non-Reactive Anti-hepatitis B virus (HBV) hepatitis B and Anti-hepatitis C antibodies (HCV) hepatitis C, Non-Reactive Human immunodeficiency virus (HIV) test, Negative Venereal Disease Research Laboratory (VDRL) test with maximum 3 months validity and allowed variation of +/-10% of the normal range
* Electrocardiogram (ECG) with no more than three months validity and with no clinically significant findings
* Pregnancy test, drug abuse test and alcohol test with negative results at selection visit and approximately 12 h before drug product administration in both study periods

Exclusion Criteria:

* Participants with some alteration in their vital signs; who fail to comply with the proposed inclusion criteria
* Participants with a history of suffering cardiovascular, renal, hepatic, muscle, metabolic, gastrointestinal, neurological problems, endocrine, hematopoietic or any type of anemia, asthma, mental illness or other organic abnormalities. Participants who have had a muscle injury within the 21 days prior to the study
* Clinically significant abnormalities in the ECG, dyspepsia, gastritis, esophagitis, gastric or duodenal ulcer; participants who require any drug product other than test product during the course of study
* Exposed to inductors or liver enzyme inhibitors or drugs capable of altering urinary pH or any potentially toxic drugs, vitamins, herbal remedies within the 30 days prior to the beginning of the study
* Participant hospitalized for any problem during the seven months prior to the study start; received investigational product within 90 days prior to the study
* Allergic to any drug product, food or substance, require special diet; positive drug abuse, alcohol, pregnancy test, breast feeding women
* Donated or lost 450 milliliter (mL) or more blood within the 60 days prior to the beginning of the study
* Participants who have not been recorded in the the Federal Commission for the Protection against Sanitary Risks (COFEPRIS) page
* Ingested alcohol, carbonated beverage, products containing xanthines, charcoal grilled nourishment, grapefruit or orange or who have smoked 24 h prior to the beginning of both study periods
* Subordination relationship between participants and investigators, an employee of the sponsor or the study site or members of their immediate family

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-08-01; Primary Completion 2015-08-01 (Actual); Study Completion 2015-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done in one center in Mexico.
Pre-assignment Details: Fifty two participants were screened for this study, out of which 15 participants were considered screening failure, 9 were kept as backup and 28 participants were randomized and all 28 of them completed the study.
Groups:
- Tylenol® Caplets (Reference), Then Mejoral® 500 Tablets (Test): Participants first received one tablet of Tylenol® Caplets [500 milligram (mg) of paracetamol], orally with 250 mL of water at room temperature, in a single dose, under minimum 10 h of fasting. After a washout period of 72 h, they then received one tablet of Mejoral® 500 tablets (500 mg of paracetamol), orally with 250 mL of water at room temperature, in a single dose, under minimum 10 h of fasting.
- Mejoral® 500 Tablets (Test), Then Tylenol® Caplets (Reference): Participants first received one tablet of Mejoral® Tablets (500 mg of paracetamol), orally with 250 ml of water at room temperature, in a single dose, under minimum 10 h of fasting. After a washout period of 72 h, they then received one tablet of Tylenol® 500 Caplets (500 mg of paracetamol), orally with 250 ml of water at room temperature, in a single dose, under minimum 10 h of fasting.
Period: Period 1
Arm/Group | Tylenol® Caplets (Reference), Then Mejoral® 500 Tablets (Test) | Mejoral® 500 Tablets (Test), Then Tylenol® Caplets (Reference)
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Washout
Arm/Group | Tylenol® Caplets (Reference), Then Mejoral® 500 Tablets (Test) | Mejoral® 500 Tablets (Test), Then Tylenol® Caplets (Reference)
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Tylenol® Caplets (Reference), Then Mejoral® 500 Tablets (Test) | Mejoral® 500 Tablets (Test), Then Tylenol® Caplets (Reference)
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: Total number of participants who were randomized and received treatment.
Arm/Group | Overall Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Last Sampling Time [AUC(0-t)]
Description: AUC(0-t) of paracetamol was calculated using the trapezoidal rule. Blood samples were taken before the administration of the reference/test product (pre-dose) and at 0.250, 0.333, 0.500, 0.667, 0.833, 1.000, 1.250, 1.500, 1.750, 2.000, 4.000, 6.000, 8.000, 12.000 and 16.000 hours (h) after each period.
Time Frame: 2 days
Population: One participant had a positive pre-dose sample in the second period of the study, equivalent to 7.74% of their Cmax, therefore, his data was not taken into account in the bioequivalence analysis
Measure: Mean (Standard Deviation); unit: hours*microgram/millilitre (h*μg/mL)
Groups:
- Tylenol® Caplets (Reference): Participants were orally administered with one caplet of Tylenol® Caplets (500 mg of paracetamol) with 250 mL of water at room temperature, in a single dose, after minimum 10 h of fasting
- Mejoral® 500 Tablets (Test): Participants were orally administered with one tablet of Mejoral® Caplets (500 mg of paracetamol) with 250 mL of water at room temperature, in a single dose, after minimum 10 h of fasting
Arm/Group | Tylenol® Caplets (Reference) | Mejoral® 500 Tablets (Test)
Number analyzed (Participants) | 27 | 27
hours*microgram/millilitre (h*μg/mL) | 15.212 (4.141) | 14.698 (4.520)
Statistical Analysis 1: Comparison: Tylenol® Caplets (Reference) vs Mejoral® 500 Tablets (Test); Test type: Non-Inferiority or Equivalence — Log-transformed PK parameter was compared between products using a linear mixed effects model including terms for product, period, sequence as fixed effect and subject nested within sequence as random effect. Bioequivalence was concluded, when the 90% confidence interval (CI) for the geometric LS mean ratios were fully contained within the predefined equivalence limits of 0.80 to 1.25; ANOVA; Ratio of Averages of Tylenol/Mejoral = 94.704, 90% CI 2-sided [88.329 to 101.540]

2. Primary Outcome: Area Under the Curve From Time Zero Extrapolated to Infinity [AUC(0-inf)]
Description: AUC(0-inf) of paracetamol was calculated using the trapezoidal rule. Blood samples were taken before the administration of the reference/test product (pre-dose) and at 0.250, 0.333, 0.500, 0.667, 0.833, 1.000, 1.250, 1.500, 1.750, 2.000, 4.000, 6.000, 8.000, 12.000 and 16.000 h after each period.
Time Frame: 2 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*μg/mL
Groups:
- Tylenol® Caplets: Participants were orally administered with one caplet of Tylenol® Caplets (500 mg of paracetamol) with 250 mL of water at room temperature, in a single dose, after minimum 10 h of fasting
- Mejoral® 500 Tablets: Participants were orally administered with one tablet of Mejoral® Caplets (500 mg of paracetamol) with 250 mL of water at room temperature, in a single dose, after minimum 10 h of fasting
Arm/Group | Tylenol® Caplets | Mejoral® 500 Tablets
Number analyzed (Participants) | 27 | 27
h*μg/mL | 15.972 (4.239) | 15.620 (4.681)
Statistical Analysis 1: Comparison: Tylenol® Caplets vs Mejoral® 500 Tablets; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of Averages of Tylenol/Mejoral = 95.989, 90% CI 2-sided [89.826 to 102.574]

3. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Cmax of paracetamol was obtained graphically from the plasma concentration over time profile. Blood samples were taken before the administration of the reference/test product (pre-dose) and at 0.250, 0.333, 0.500, 0.667, 0.833, 1.000, 1.250, 1.500, 1.750, 2.000, 4.000, 6.000, 8.000, 12.000 and 16.000 h after each period.
Time Frame: 2 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micogram per mililitre (μg/mL)
Arm/Group | Tylenol® Caplets | Mejoral® 500 Tablets
Number analyzed (Participants) | 27 | 27
micogram per mililitre (μg/mL) | 7.182 (2.841) | 8.118 (3.938)
Statistical Analysis 1: Comparison: Tylenol® Caplets vs Mejoral® 500 Tablets; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of Averages of Tylenol/Mejoral = 106.132, 90% CI 2-sided [85.151 to 132.283]

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Tmax of paracetamol was obtained graphically from the plasma concentration over time profile. Blood samples were taken before the administration of the reference/test product (pre-dose) and at 0.250, 0.333, 0.500, 0.667, 0.833, 1.000, 1.250, 1.500, 1.750, 2.000, 4.000, 6.000, 8.000, 12.000 and 16.000 h after each period.
Time Frame: 2 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours (h)
Arm/Group | Tylenol® Caplets | Mejoral® 500 Tablets
Number analyzed (Participants) | 27 | 27
Hours (h) | 0.719 (0.474) | 0.738 (0.501)

ADVERSE EVENTS:
Time Frame: upto 14 days after administration of investigational product
Description: MedDRA
Groups:
- Tylenol® Caplets: Participants will first receive one tablet [500 milligram (mg) of paracetamol] of Tylenol® Caplets, orally with 250 mL of water at room temperature, in a single dose, under minimum 10 h fasting. After a washout period of 72 h, they then will receive one tablet (500 mg of paracetamol) of Mejoral® 500 tablets, orally with 250 mL of water at room temperature, in a single dose, under minimum 10 h fasting.
- Mejoral® 500 Tablets: Participants will first receive one tablet (500 mg of paracetamol) of Mejoral® 500 tablets, orally with 250 mL of water at room temperature, in a single dose, under minimum 10 h fasting. After a washout period of 72 h, they then will receive one tablet (500 mg of paracetamol) of Tylenol® Caplets, orally with 250 mL of water at room temperature, in a single dose, under minimum 10 h fasting.
Arm/Group | Tylenol® Caplets | Mejoral® 500 Tablets
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.